CLINICAL TRIAL: NCT03993054
Title: Web-Based Cognitive Behavioral Stress Management for Latino Sexual Minority Men Living With HIV and Cancer
Acronym: C-SmartManage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sara StGeorge, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200127; U54MD002266 (NIH)
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Results first posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: HIV/AIDS; Cancer
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally-tailored CBSM (Experimental): Participants will receive web-based CBSM that is culturally-tailored for Latino men specifically over 10 weeks.
  Interventions: Behavioral: Culturally-tailored cognitive behavioral stress management

INTERVENTIONS:
Behavioral: Culturally-tailored cognitive behavioral stress management — The SmartManage CBSM intervention includes content that is of clinical relevance to sexual minority men dually diagnosed with HIV and cancer. Intervention content includes: co-management of HIV and cancer, strategies for self-advocacy, partnering with the health system and health providers, intimacy and disclosure concerns regarding both conditions, and contextual stressors (e.g., racial/ethnic minority status), stigmatization, assertiveness and communication skills, and self-efficacy in care coordination. Participants receive weekly 1.5 hour interactive group sessions online that focus on stress and self-management skill-building, and also receive access to didactic information regarding intervention content via the intervention website. Intervention length is 10 weeks. This intervention will be a version of SmartManage that is culturally-tailored for Latino populations.
  Other Names: C-SmartManage

SUMMARY:
This is a one year study to develop and test a culturally-tailored, web-based cognitive behavioral stress management (CBSM) intervention for Latino sexual minority men living with both HIV and cancer. Sexual minority Latino men living with HIV and cancer experience a variety of health disparities related to their diagnoses, including higher distress. The project will use a single-group pre-post design. The project will use a community-based participatory research approach, and the investigators have included (and will continue to include) LGBT-serving community partners in all phases of the research from study design to implementation and dissemination of findings. The proposed study will aid in attenuating health disparities among Latino sexual minority men living with HIV and cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with at least one form of non-metastatic solid tumor cancer,
2. Are ≥ 30 days post active primary treatment (i.e. surgery, radiation, and/or chemotherapy*) for their cancer. (Note: Adjuvant therapies, such as hormone therapy for prostate cancer, etc. are not considered exclusionary),
3. Self-identify as a sexual minority man,
4. have been diagnosed with HIV,
5. Have reliable access to a computer/device with internet accessibility, and
6. Are fluent English.

Exclusion Criteria:

1. Have had one of the following exclusionary cancer types: Leukemia (or other cancers of the blood), Non-melanoma skin cancer only (not in combination with another type listed in the inclusion criteria above), Brain cancer, Eye cancer, a form of pediatric cancer (if the pediatric cancer is the only cancer diagnosis the patient has had),
2. Have a history of advanced (metastatic) cancer of any type or are currently undergoing primary treatment for their cancer,
3. Have had inpatient treatment for severe mental illness in the past 12 months, or have overt signs of psychopathology (i.e. psychosis) and/or suicidality at the time of screening,
4. Are experiencing active alcohol dependence, or have had inpatient treatment for alcohol abuse within the past 12 months,
5. Are experiencing active substance dependence, or have had inpatient treatment for substance abuse within the past 12 months, and/or
6. Have any other medical conditions resulting in a predicted life expectancy <12 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender males
Enrollment: 16 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara St. George, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixteen adults signed informed consent form and were allocated to the intervention. PI removed one from the study for providing false information.
Period: Overall Study
Arm/Group | Culturally-tailored CBSM
Started | 16
Completed | 15
Not Completed | 1
Not completed — PI Decision | 1

BASELINE CHARACTERISTICS:
Population: Sixteen adults signed an informed consent form and were allocated to the intervention. The principal investigator removed one participant from the study and its analysis for providing false information.
Arm/Group | Culturally-tailored CBSM
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 2
  Unknown or Not Reported | 2
General Stress [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale (PSS) consists of 10 items, which are summed to create a total score ranging from 0 to 40. Higher scores indicate greater levels of perceived stress.
  units on a scale | 31.7 (8.4)
Disease-Related Distress [Mean (Standard Deviation); unit: units on a scale] — The Impact of Events Scale-Revised (IES-R) measures the psychological impact of traumatic events. It consists of three subscales: intrusion (eight items), avoidance (eight items), and hyperarousal (six items). Each subscale score is calculated by summing the items within that subscale. The maximum possible score for intrusion and avoidance is 32 each, while hyperarousal has a maximum score of 24. The scores from these subscales are summed to create a total score, which ranges from 0 to 88. Higher scores indicate a greater negative impact of the traumatic event.
  units on a scale
    Intrusion | 11.7 (7.3)
    Avoidance | 12.9 (6.7)
    Hyperarousal | 8.0 (6.0)
    Total Score | 32.6 (18.2)
Health Related Quality of Life (FACT-G) [Mean (Standard Deviation); unit: units on a scale] — The Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire was used to assess quality of life. It comprises four sub-scales: physical well-being (7 items, score range 0-28), social/family well-being (7 items, score range 0-28), emotional well-being (6 items, score range 0-24), and functional well-being (7 items, score range 0-28). The overall score is calculated by summing the scores of these four sub-scales, resulting in a total possible score range of 0-108. Higher scores on the FACT-G indicate a better quality of life.
  units on a scale
    Physical Well-being | 20.3 (6.5)
    Social Well-being | 16.1 (6.8)
    Emotional Well-being | 15.5 (4.2)
    Functional Well-being | 16.9 (6.4)
    Total Score | 68.9 (15.7)
Health Related Quality of Life (MOS-HIV) [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study HIV Survey (MOS-HIV) assesses 10 health dimensions (i.e., health perceptions, pain, physical functioning, role functioning, social functioning, cognitive functioning, mental health, energy, health distress, and quality of life). Subscales are scored on a 0-100 scale, with a higher score indicating better health.
  units on a scale
    Pain | 8.5 (2.3)
    Physical Functioning | 13.7 (3.7)
    Social Functioning | 4.4 (1.7)
    Role Functioning | 2.7 (1.1)
    Mental Health | 19.9 (3.9)
    Health Distress | 17.3 (5.0)
    Cognitive Functioning | 17.9 (5.2)
    Vitality/Energy | 13.8 (3.6)
    General Health | 14.4 (5.4)
    Health Perception | 3.2 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in General Stress
Description: The Perceived Stress Scale (PSS) consists of 10 items, which are summed to create a total score ranging from 0 to 40. Higher scores indicate greater levels of perceived stress. The outcome was analyzed as the change from baseline.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Culturally-tailored CBSM
Number analyzed (Participants) | 15
units on a scale | -1.8 (10)

2. Primary Outcome: Change in Disease-Related Distress
Description: The Impact of Events Scale-Revised (IES-R) measures the psychological impact of traumatic events. It consists of three subscales: intrusion (eight items), avoidance (eight items), and hyperarousal (six items). Each subscale score is calculated by summing the items within that subscale. The maximum possible score for intrusion and avoidance is 32 each, while hyperarousal has a maximum score of 24. The scores from these subscales are summed to create a total score, which ranges from 0 to 88. Higher scores indicate a greater negative impact of the traumatic event. The outcome was analyzed as the change from baseline.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Culturally-tailored CBSM
Number analyzed (Participants) | 15
units on a scale
  Intrusion | -3.2 (6.4)
  Avoidance | -5.0 (7.2)
  Hyperarousal | -1.9 (6.2)
  Total Score | -10.2 (17.8)

3. Primary Outcome: Change in Health-Related Quality of Life (FACT-G)
Description: The Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire was used to assess quality of life. It comprises four sub-scales: physical well-being (7 items, score range 0-28), social/family well-being (7 items, score range 0-28), emotional well-being (6 items, score range 0-24), and functional well-being (7 items, score range 0-28). The overall score is calculated by summing the scores of these four sub-scales, resulting in a total possible score range of 0-108. Higher scores on the FACT-G indicate a better quality of life. The outcome was analyzed as the change from baseline.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Culturally-tailored CBSM
Number analyzed (Participants) | 15
units on a scale
  Physical Well-being | -1.5 (8)
  Social Well-being | 0.2 (4.3)
  Emotional Well-being | 3.5 (3.8)
  Functional Well-being | 0.4 (3.9)
  Total Score | 2.7 (12.1)

4. Primary Outcome: Change in Health-Related Quality of Life (MOS-HIV)
Description: The Medical Outcomes Study HIV Survey (MOS-HIV) assesses 10 health dimensions (i.e., health perceptions, pain, physical functioning, role functioning, social functioning, cognitive functioning, mental health, energy, health distress, and quality of life). Subscales are scored on a 0-100 scale, with a higher score indicating better health. The outcome was analyzed as the change from baseline.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Culturally-tailored CBSM
Number analyzed (Participants) | 15
units on a scale
  Pain | -1 (2.4)
  Physical Functioning | -0.2 (4.7)
  Social Functioning | -0.2 (2.5)
  Role Functioning | 0.6 (0.8)
  Mental Health | 0.7 (6.3)
  Health Distress | -2.5 (8.5)
  Cognitive Functioning | -1.3 (6.3)
  Vitality/Energy | -0.8 (3.8)
  General Health | 0.8 (5)
  Health Perception | 0.3 (0.8)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Culturally-tailored CBSM
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03993054/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03993054/ICF_001.pdf